CLINICAL TRIAL: NCT06142279
Title: Development and Qualification of Methods for Analyzing the Mucosal Immune Response to COVID-19
Acronym: MUCOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DR230062-MUCOVID
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Certain Disorders Involving the Immune Mechanism
MeSH Terms: interventions — Polymerase Chain Reaction

STUDY DESIGN:
Intervention Model Description: Multicenter cross-sectional study comparing short-term mucosal response in individuals recently infected with SARS-CoV-2 versus recently non-infected individuals. The study will consist of two parts:
  1. Part A, which focuses on developing the technique, involves prospective data collection and the collection of biological samples (nasal, salivary, and blood samples).
  2. Part B, which aims to qualify the analysis method, also includes prospective data collection and the collection of biological samples.
  Once the threshold is reached in one of the two groups in Phase A, Phase B will begin concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID + (Other): participant with a positive SARS-CoV-2 PCR test
  Interventions: Biological: Sampling; Biological: PCR (polymerase chain reaction) SARS-CoV-2
- COVID - (Other): participant with a negative SARS-CoV-2 PCR test
  Interventions: Biological: Sampling; Biological: PCR (polymerase chain reaction) SARS-CoV-2

INTERVENTIONS:
Biological: Sampling — At baseline, nasal, salivary and blood sampling will be taken for the participants.
Biological: PCR (polymerase chain reaction) SARS-CoV-2 — At baseline, this PCR SARS-CoV-2 will be taken for the participants.

SUMMARY:
The pandemic associated with the SARS-CoV-2 coronavirus has affected over 760 million individuals worldwide, resulting in more than 6.9 million deaths. France has also been heavily impacted, with over 39.8 million infections and 167,000 deaths.

SARS-CoV-2 primarily causes an upper respiratory tract infection transmitted through the air. When it reaches the lungs, it leads to a severe acute respiratory illness called COVID-19. The body's response to this viral assault primarily occurs at the level of the respiratory mucosa.

This mucosal response is complex, involving various levels of activity. Mucosal immunity is therefore essential for an adequate and long-term immune response against viral respiratory infections, including SARS-CoV-2 infection.

Infection with SARS-CoV-2 triggers a humoral immune response with the production of antibodies in the blood (serum antibodies) and antibodies in the upper respiratory tract (mucosal antibodies). It also induces a cellular immune response by activating specific blood T lymphocytes.

Tests used to measure the humoral blood response against SARS-CoV-2 and their neutralizing capacity are now well identified, as are tests for assessing the serum cellular T lymphocyte response. However, tests for measuring mucosal immune responses are not routinely used.

Our study aims to develop and qualify methods for analyzing mucosal immunity directed against SARS-CoV-2. These methods will be essential for a more precise analysis of the body's mucosal response to this virus.

Once these analytical methods are validated, they will enable the study of mucosal responses to infection, as well as mucosal responses induced by vaccination against SARS-CoV-2, particularly in the context of future nasal vaccine use.

DETAILED DESCRIPTION:
SARS-CoV-2 is initially responsible for an airborne infection of the upper respiratory tract which, on reaching the lungs, causes a severe acute respiratory illness known as COVID-19.

The organism's response to this viral aggression is initially directed at the respiratory mucosa.

This mucosal response is complex, with different levels of activity interacting: mechanical activity, with the secretion of mucus that acts as a barrier to the infectious agent; physico-chemical activity, with the production of enzymes and cytokines that contribute to the degradation of viral particles; and specific humoral immune activity, with the production of secretory IgA-type immunoglobulins at the mucosal level, with neutralizing activity that blocks viral entry into the host cell.

These innate and adaptive immune mechanisms, together with their humoral and cellular components, play an essential role in mucosal barrier function. Mucosal immunity is therefore essential for an adequate, early and long-term immune response against respiratory viral infections.

SARS-CoV-2 is an enveloped virus with a helical capsid and a genome consisting of approximately 30,000 nucleotides. This genome codes for several proteins essential for virion formation, including the S protein for Spike and the N protein for nucleocapsid.

The viral S protein binds to the host cell's angiotensin-converting enzyme 2 (ACE2). ACE2 thus acts as a viral receptor mediating viral entry into the cell and the triggering an immune response in the host. This protein S is the main target of the neutralizing antibody response. Mutations in protein S have been responsible for the emergence of variants of SARS-CoV-2 with different phenotypes affecting transmission and susceptibility to antibody.

The N protein is a highly immunogenic glycoprotein also involved in viral replication and in the modulation of cellular signalling pathways. During virion assembly virion, the N protein binds to viral RNA and leads to the formation of the helical nucleocapsid. This N protein is highly conserved in all SARS-CoV-2 variants and may therefore be an interesting target in the universal defense against this virus.

In the event of a respiratory infection, stimulation of the mucosal immune system triggers on the one hand, a humoral response with the release of secretory immunoglobulins, mainly secretory IgA. The main role of IgA is to prevent the virus from spreading throughout the body.

On the other hand, respiratory infection will also trigger a mucosal cellular response primarily mediated by T lymphocytes.

Infection with SARS-CoV-2 triggers an immune response involving antibody production in the blood (serum antibodies), stimulation of blood lymphocytes and antibody production in the upper respiratory tract (mucosal antibodies). The quantitative anti-SARS-CoV-2 humoral response in the blood (serum antibodies) has been assessed by various tests. For the time being, however, it relies mainly on EIA-type tests, with blood levels of anti-S IgG (directed against the Spike protein) and anti-N IgG (directed against the nucleocapsid protein). Qualitative analysis of this response is based on the ability of these antibodies to have neutralizing activity (neutralizing antibodies).

The anti-SARS-CoV-2 T lymphocyte cellular response also appears to be important in controlling infection. The most rapid test for assessing this T lymphocyte response is the ELISPOT IFN-γ

As for the mucosal humoral response, several studies have documented the presence of virus-specific anti-S IgA antibodies (directed against the Spike protein) in the nasopharyngeal secretions or saliva of infected individuals. To date, there is no routinely-used test for measuring mucosal antibodies to SARS-CoV-2, notably secretory anti-S IgA, and to analyze their neutralizing activity.

Our study will thus enable us to develop and qualify methods for analyzing mucosal immunity to SARS-CoV-2. These methods will be essential for analyzing mucosal response to this virus.

Once these analytical methods have been validated, they will make it possible to study the mucosal response to infection but also the mucosal response induced by vaccination against SARS-CoV-2, particularly when using nasal vaccines.

Indeed, the vaccines currently used to combat SARS-CoV-2 induce serum neutralizing activity against protein S (Spike). Their intramuscular route of administration will induce systemic immunity, providing protection against severe forms of the infection. Nevertheless, mucosal immunity induced by current vaccines remains low. The development of a nasally-administered vaccine is an interesting avenue, as it would provide more complete protection, notably by controlling virus replication in the upper respiratory tract, thus inducing upper respiratory tract, thereby inducing herd immunity and reducing transmission of the virus.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Participant affiliated with a social security scheme
* Participant willing to take part in the study and having provided consent
* Participant in good health or with a stable chronic condition for more than 6 months

Exclusion Criteria:

* Contraindication for nasopharyngeal sampling
* Pregnant or breastfeeding women
* Participants benefiting from a legal protection measure as referred to in articles L1121-5 to L1121-8 of the Public Health Code (guardianship, trusteeship, etc.)
* Participant with an acute condition unrelated to SARS-CoV-2 infection
* Participant with an unstable chronic condition

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To study the anti-Spike mucosal humoral immune response by measuring secretory IgA in nasal secretions | Baseline - Day 0
  The level of secretory IgA (immunoglobulin A) in nasal secretions, expressed in picograms per milliliter equivalent.
Analysis of the neutralizing capacity of anti-Spike IgA in nasal secretions | Baseline - Day 0
  The neutralizing capacity of secretory nasal IgA assessed in neutralization titer (PRNT 50).

SECONDARY OUTCOMES:
Determination of secretory anti-Spike IgA in salivary secretions | Baseline - Day 0
  Secretory IgA levels in saliva expressed in picograms per milliliter Eq
Analysis of the neutralizing capacity of anti-Spike IgA in salivary secretions | Baseline - Day 0
  Salivary IgA neutralizing capacity assessed by neutralizing titer (PRNT 50)
Determination of serum anti-Spike IgG | Baseline - Day 0
  Blood anti-S IgG (immunoglobulin G) levels expressed in Binding Antibody Units per milliliter (BAU/ml)
Analysis of the neutralizing capacity of serum anti-Spike IgG | Baseline - Day 0
  Blood IgG neutralizing capacity assessed by neutralizing titer (PRNT 50)
Assay serum anti-N IgG | Baseline - Day 0
  Blood anti-N IgG levels expressed as an index
Study the systemic cellular immune response by measuring interferon-gamma production | Baseline - Day 0
  T-cell reactivity expressed in the number of Spot Forming Units per 106 Peripheral Blood Mononuclear Cells (SFU: Spot Forming Unit)

CONTACTS AND LOCATIONS:
Overall Officials: Zoha MAAKAROUN-VERMESSE, MD-PHD, Principal Investigator — CHRU de TOURS
Locations (1):
- CHRU de Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haute autorité de santé. Aspect immunologiques et virologiques de l'infection par le SARS-CoV-2 ; Rapport HAS 25 Novembre 2020
- [Background] Alu A, Chen L, Lei H, Wei Y, Tian X, Wei X. Intranasal COVID-19 vaccines: From bench to bed. EBioMedicine. 2022 Feb;76:103841. doi: 10.1016/j.ebiom.2022.103841. Epub 2022 Jan 24. PMID 35085851
- [Background] Y. Jouan · M. Si-Tahar · A. Guillon. Immunité de la muqueuse respiratoire : physiologie et implications en réanimation. Méd. Intensive Réa 2017 ; 26 :11-20
- [Background] Smith N, Goncalves P, Charbit B, Grzelak L, Beretta M, Planchais C, Bruel T, Rouilly V, Bondet V, Hadjadj J, Yatim N, Pere H, Merkling SH, Ghozlane A, Kerneis S, Rieux-Laucat F, Terrier B, Schwartz O, Mouquet H, Duffy D, Di Santo JP. Distinct systemic and mucosal immune responses during acute SARS-CoV-2 infection. Nat Immunol. 2021 Nov;22(11):1428-1439. doi: 10.1038/s41590-021-01028-7. Epub 2021 Sep 1. PMID 34471264
- [Background] Chavda VP, Vora LK, Pandya AK, Patravale VB. Intranasal vaccines for SARS-CoV-2: From challenges to potential in COVID-19 management. Drug Discov Today. 2021 Nov;26(11):2619-2636. doi: 10.1016/j.drudis.2021.07.021. Epub 2021 Jul 29. PMID 34332100
- [Background] Denis F, Alain S, Hantz S, Lagrange P. [Antiviral vaccination and respiratory mucosal immunity: still disappointing results from a seductive idea]. Presse Med. 2005 Oct 8;34(17):1245-53. doi: 10.1016/s0755-4982(05)84165-x. French. PMID 16230967
- [Background] Russell MW, Mestecky J. Mucosal immunity: The missing link in comprehending SARS-CoV-2 infection and transmission. Front Immunol. 2022 Aug 17;13:957107. doi: 10.3389/fimmu.2022.957107. eCollection 2022. PMID 36059541
- [Background] Tang J, Zeng C, Cox TM, Li C, Son YM, Cheon IS, Wu Y, Behl S, Taylor JJ, Chakaraborty R, Johnson AJ, Shiavo DN, Utz JP, Reisenauer JS, Midthun DE, Mullon JJ, Edell ES, Alameh MG, Borish L, Teague WG, Kaplan MH, Weissman D, Kern R, Hu H, Vassallo R, Liu SL, Sun J. Respiratory mucosal immunity against SARS-CoV-2 after mRNA vaccination. Sci Immunol. 2022 Oct 28;7(76):eadd4853. doi: 10.1126/sciimmunol.add4853. Epub 2022 Oct 21. PMID 35857583
- [Background] Yaugel-Novoa M, Bourlet T, Paul S. Role of the humoral immune response during COVID-19: guilty or not guilty? Mucosal Immunol. 2022 Jun;15(6):1170-1180. doi: 10.1038/s41385-022-00569-w. Epub 2022 Oct 4. PMID 36195658